CLINICAL TRIAL: NCT01097876
Title: A Phase 1, Double-Blind, Placebo-Controlled, Sponsor Open, Randomized, Multiple Dose Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-04447943 In Healthy Volunteers When Combined With Donepezil
Brief Title: A Study To Evaluate The Safety, Tolerability And Plasma Drug Levels Of PF-04447943 When Administered With Donepezil To Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B0401012
Record Dates: First submitted 2010-03-23; First posted 2010-04-02 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: healthy volunteer; pharmacokinetic; safety
MeSH Terms: interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active PF-04447943 (Experimental)
  Interventions: Drug: PF-04447943 25 mg
- Placebo PF-04447943 (Placebo Comparator)
  Interventions: Drug: Placebo PF

INTERVENTIONS:
Drug: PF-04447943 25 mg — 25 mg PF-04447943 BID for 7 days (period 1) 7 day washout (no drug) 7 days of 5 mg donepezil QD; 14 days 10 mg QD (Period 2) 7 days of 10 mg donepezil QD and 25 mg PF-04447943 BID (Period 3)
  Arms: Active PF-04447943
Drug: Placebo PF — Placebo BID for 7 days (period 1) 7 day washout (no drug) 7 days of 5 mg donepezil QD; 14 days 10 mg QD (Period 2) 7 days of 10 mg donepezil QD and Placebo BID (Period 3)
  Arms: Placebo PF-04447943

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of PF-04447943, before and after multiple doses of donepezil in healthy volunteers. Evaluate the plasma drug levels of both PF-04447943 and donepezil.

DETAILED DESCRIPTION:
Evaluate the safety and tolerability of PF-04447943, before and after multiple doses of donepezil in healthy volunteers. Evaluate the plasma drug levels of both PF-04447943 and donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential subjects between the ages of 21 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing females; females of childbearing potential.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Steady state PF 04447943 Cmax and AUCtau. | up through day 44
Steady state Donepezil Cmax and AUCtau. | up through day 44
Safety endpoints include vital signs, ECGs, clinical laboratory tests, clinical examinations, and adverse events. | up through day 44

SECONDARY OUTCOMES:
There are no Secondary Endpoints | There are no Secondary Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401012&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Plasma%20Drug%20Levels%20Of%20PF-04447943%20When%20Administered%20With%20Donepezil%20To%20Healthy%20Volunte